CLINICAL TRIAL: NCT05020756
Title: A Retrospective Study in Children Who Have Switched to Isosource Junior Mix Formula (RICIMIX Study)
Brief Title: Study in Children Who Have Switched to Isosource Junior Mix Formula
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Blend 002
Record Dates: First submitted 2021-04-28; First posted 2021-08-25 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Dietary Supplement: Isosource Junior Mix — Single arm study, collecting data on those who have been on Isosourcr Junior mix tube feed formula for 30 days

SUMMARY:
A Retrospective study In Children who have switched to Isosource Junior Mix formula (RICIMIX study) will review paediatric children > 12 months of age who require Isosource Junior Mix as an enteral tube feeding formula and have consumed the formula for at least 1 month. The purpose of this study is to understand If there has been an improvement in outcomes/ experiences

* The current usage of ISJMIX formula in children who require blended diets
* Improved feeding intolerances
* Improved patient outcomes/ experiences

DETAILED DESCRIPTION:
Retrospective data will be collected using questionnaire by the dietitians at the nutrition and dietetic department. All completed questionnaires will be sent back to Nestle Health Science/ CRO company.

The primary objectives:

The following measures will be collected retrospectively after 1 month use of ISJMIX

* Feeding tolerance [no change, tolerance improved, tolerance worsened]: gastric residuals, gagging/retching, vomiting, abdominal distention/ gas, stool consistency issues (too hard, too loose)
* Volume of formula consumed in a day

The secondary objective is to collect restropective data on:

* Any improved patient outcomes noted
* Calculate the potential cost savings made when using ISJMIX to help manage the feeding intolerances
* Calculate the potential costs benefit of using ISJMIX over other standard formulas

ELIGIBILITY:
Inclusion Criteria:

* All children who are using Isosource Junior Mix as tube feed formula

Exclusion Criteria:

* All children who did not switch to Isosource Junior Mix feed formula

Ages: 12 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatric children > 12 months of age who require Isosource Junior Mix as an enteral tube feeding formula and have consumed the formula for at least 1 month
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Feeding tolerance | 30 days
  The following measures will be collected retrospectively after 1 month use of ISJMIX
  • Feeding tolerance [no change, tolerance improved, tolerance worsened]: gastric residuals, gagging/retching, vomiting, abdominal distention/ gas, stool consistency issues (too hard, too loose)

SECONDARY OUTCOMES:
Volume consumed | 30 days
  Average volume consumed over month period
Weight in Kg | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Nestle Health Science, Gatwick, United Kingdom

IPD SHARING:
Plan to Share IPD: No